CLINICAL TRIAL: NCT06880328
Title: 18F-Dihydroxyphenylalanine (DOPA) Positron Emission Tomography (PET), Randomized, Double-blind, Crossover Study to Explore Dopamine Synthesis Capacity in the Whole Striatum After 2 Weeks of Treatment With 150mg of RO6889450 or Placebo in Patients With Schizophrenia
Brief Title: 18F-Dihydroxyphenylalanine (DOPA) Positron Emission Tomography (PET) Study to Explore Dopamine Synthesis Capacity in the Whole Striatum After 2 Weeks of Treatment With Ralmitaront or Placebo in Participants With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BP39833
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — fluorodopa F 18

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence 1: Ralmitaront then Placebo (Experimental): Participants were given a daily dose of Ralmitaront during the treatment period of 14 days, followed by a 7 day washout period, and then a daily dose for 14 days with the placebo.
  Interventions: Drug: Ralmitaront; Other: Radiolabeled PET tracer [18F]-DOPA; Drug: Placebo
- Sequence 2: Placebo then Ralmitaront (Experimental): Participants were given a daily dose of the placebo during the 14 day period, followed by a 7 day washout, and then a daily dose of Ralmitaront for 14 days.
  Interventions: Drug: Ralmitaront; Other: Radiolabeled PET tracer [18F]-DOPA; Drug: Placebo

INTERVENTIONS:
Drug: Ralmitaront — Participants were given a once 150 mg daily dose of Ralmitaront orally during the 14 day treatment period.
  Other Names: RO6889450
Other: Radiolabeled PET tracer [18F]-DOPA — [18 F]-DOPA solution for injection is manufactured by the PET imaging centers according to specifications established for the tracer at the site. The injection will happen prior to the scan being done and will last for approximately 30 seconds.
Drug: Placebo — Participants were given a daily dose of the placebo during the 14 day treatment period.

SUMMARY:
This study is an exploratory proof of mechanism (POM) study using PET/functional magnetic resonance imaging (fMRI) in a 2-period, 2-sequence, crossover design. The aim of the study is to confirm the potential of Ralmitaront to decrease dopamine synthesis capacity (DSC) - as measured by levels of F-DOPA - in the striatum of participants with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Male patients with non-acute schizophrenia defined by DSM-5 diagnosis of schizophrenia as established by the mini-international neuropsychiatric interview (MINI)
* Medically stable over 1 month and psychiatrically stable for at least 3 months prior to the screening visit
* Patients with evidence of clear treatment response to antipsychotics as documented by chart information or reported by the patient or an informant considered reliable by the Investigator
* Outpatient with no hospitalization for worsening of schizophrenia within 3 months prior to screening (hospitalization for social management within this time was acceptable)
* At least one positive and negative syndrome scale (PANSS) positive subscale item from P1 (delusion), P3 (hallucination), P5 (grandiosity), or P6 (suspiciousness/persecution) of mild or greater severity (score .3), but below 7 (extreme severity)
* Body mass index (BMI) between 18 and 35 kg/m2 inclusive

Exclusion Criteria:

* Diagnosis for bipolar disorder, schizoaffective disorder or major depressive disorder based on DSM-5
* A prior or current general medical condition that might be impairing central nervous system (CNS) functioning (e.g., head trauma with persistent clinically significant neurological or cognitive sequelae, dementia, seizure disorder, stroke, neurodegenerative, inflammatory, infectious, neoplastic, toxic, metabolic or endocrine disorders)
* Average triplicate QTcF interval greater than 450 msec or other clinically significant abnormality on screening electrocardiogram (ECG) as assessed by the Investigator or deputy based on centralized reading
* Clinically significant abnormalities in laboratory safety test results (including hepatic and renal panels, complete blood count, chemistry panel and urinalysis)
* Positive result at screening for hepatitis B (HBV), hepatitis C (HCV, untreated), or human immunodeficiency virus (HIV)-1 and HIV-2. HCV patients who had been successfully treated and who tested negative for HCV ribonucleic acid (RNA), could be considered eligible for entry into the study
* Patient at current significant risk of suicide or harming him or others according to the Investigator's judgment
* Patients with a history of violent/suicidal/homicidal behavior or history of suicidal/homicidal command hallucinations in the past 10 years
* Patients who have had 3 or more exacerbations associated with violent/suicidal/homicidal behavior or suicidal/homicidal command hallucinations (regardless of time)
* History of electroconvulsive treatment (ECT)
* Patients treated with long-acting injectable antipsychotic drugs or cariprazine
* Patients with known history of treatment resistance or having received clozapine within 3 months of screening
* Treatment with prohibited medication taken within 4 weeks (or within 5 times the elimination half-life of the medication) before the first study drug administration (whichever is longer). This included medications with known effects on cerebral blood flow.
* Use of grapefruit, Seville orange or star fruit containing products within 1 week before the first study drug administration
* Receipt of an investigational drug within 90 days or 5 times the half-life of the investigational drug, whatever was longer, prior to baseline visit
* Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per Investigator assessment)
* Moderate-to-severe substance use disorder within 6 months of screening (excluding caffeine) as defined by DSM-5
* Heavy smokers as defined by a high dependence score in the Fagerstrom Tolerance Scale (score ≥ 6)
* Positive urine drug screen for amphetamines, methamphetamines, opiates, buprenorphine, methadone, cannabinoids, cocaine and barbiturates after informed consent and prior to randomization
* Any sensorial impairment such as deafness and reduced visual acuity, which could not be corrected in the MRI scanner
* Clinically significant abnormal findings on the baseline MRI images such as stroke, infarction, space-occupying lesion such as tumor, structural abnormalities, or vascular pathology
* Known exposure to radiation in the last year that would mean the total exposure to radiation with participation in the study was likely to exceed 30 mSv
* Donation of blood over 400 mL within 3 months prior to screening

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2019-09-04 (Actual); Study Completion 2019-09-04 (Actual)

PRIMARY OUTCOMES:
Influx Rate Constant (Ki) Value of [18F]-DOPA in the Whole Striatum, as Measured Using [18F]-DOPA PET Imaging | Baseline, and on Days 13-14 and Days 34-35

SECONDARY OUTCOMES:
Bilateral Ventral Striatum Eigenvariates From the T-Contrast of Rewarded vs. Non-reward Expectation During the Monetary Incentive Delay (MID) Task, as Assessed Using fMRI | Baseline, and on Days 13-14 and Days 34-35
Percentage of High Effort Choices Under Deterministic Reward Condition for High Reward in the Effort-Choice Benefit Task | Baseline, and on Days 13-14 and Days 34-35
Mean Cerebral Blood Flow (CBF) in Different Brain Regions, as Measured by fMRI | Baseline, and on Days 13-14 and Days 34-35
Bilateral Eigenvariate From Dorsolateral Prefrontal Regions Defined Based on the 2-back >0-back Contrast in the N-back Working Memory Task, as Assessed Using fMRI | Baseline, and on Days 13-14 and Days 34-35
Incidence and Severity of Adverse Events (AEs) | From first dose until 14 days after the last dose of study treatment (up to 49 days)
Incidence of Treatment Discontinuations Due to AEs | From first dose until 14 days after the last dose of study treatment (up to 49 days)
Incidence of Vitals Sign Abnormalities (Resting and Orthostatic) | From first dose until 14 days after the last dose of study treatment (up to 49 days)
Change From Baseline in ECG Intervals: PQ (PR), QRS, QT, RR and QTcF | Baseline, Days 13-14, 21, 34-35, and during the follow-up visit (14-18 days after last dose)
Incidence of Laboratory Abnormalities, Based on Hematology, Clinical Chemistry, and Urinalysis Test Results | From first dose until 14 days after the last dose of study treatment (up to 49 days)
Concentration of Ralmitaront and Ralmitaront-derived Metabolite(s) Per Time-point | Days 2, 7, 13-14, 23, 28, 34-35, and during the follow up visit (14-18 days after last dose)
Area Under the Curve (AUCss) of Ralmitaront and Ralmitaront-derived Metabolite(s) | Days 2, 7, 13-14, 23, 28, 34-35, and during the follow up visit (14-18 days after last dose)
Cmax of Ralmitaront and Ralmitaront-derived Metabolite(s) | Days 2, 7, 13-14, 23, 28, 34-35, and during the follow up visit (14-18 days after last dose)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- United States (4):
  - Parexel California Clinical Trials Medical Group, Glendale, California
  - Collaborative Neuroscience Network Inc., Torrance, California
  - CBH Health, Gaithersburg, Maryland
  - St Louis Clinical Trials, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No